CLINICAL TRIAL: NCT00790868
Title: Exposure, D-Cycloserine Enhancement, and Genetic Modulators in Panic Disorder
Acronym: DCSPanic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Otto, Ph.D., Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH081116 (NIH); R01MH081116 (NIH)
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Panic Disorder
Keywords: Panic Disorder; Anxiety; D-cycloserine; DCS; Cognitive Behavioral Therapy; CBT
MeSH Terms: conditions — Panic Disorder; Anxiety Disorders | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- D-cycloserine (Experimental): DCS-augmented CBT
  Interventions: Drug: d-cycloserine
- Placebo (Placebo Comparator): placebo-augmented CBT
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: d-cycloserine — 50mg
  Other Names: DCS
  Arms: D-cycloserine
Drug: placebo — 50mg
  Arms: Placebo

SUMMARY:
This is a 5-year double blind, randomized, controlled, trial conducted at three treatment sites, aimed at showing the acute and longer-term effects of DCS augmentation of exposure-based CBT for panic disorder relative to placebo augmentation. By demonstrating that DCS can enhance the results of even a brief treatment strategy, the investigators are seeking to validate an approach that fits well with the practice limitations and applications of CBT in effectiveness studies.

DETAILED DESCRIPTION:
In this application, the investigators propose to further validate and expand upon one of the apparent striking successes of translational research. Specifically, basic research on the neural circuitry underlying fear extinction led to the examination of d-cycloserine (DCS), a partial agonist of the NMDA receptor in the amygdala, as an agent capable of enhancing extinction learning (Davis et al., 2006; Davis et al., in press). Following successful validation of this strategy in the animal laboratory (see Ledgerwood et al., 2005; Richardson et al., 2004), Ressler et al. (2004) showed that single doses of d-cycloserine (DCS) could enhance extinction in a human exposure paradigm for height phobic adults. This exciting initial finding was replicated by this research team for the treatment of social anxiety disorder (Hofmann et al., 2006), as well as an initial pilot study of the treatment of panic disorder (Tolin et al., 2006). As discussed by Anderson and Insel (2006), these findings have the potential to foster significant advances in the treatment of anxiety disorders. The present study represents the further application of DCS for augmenting the effects of exposure-based cognitive-behavior therapy (CBT), now applied to the treatment of panic disorder with or without agoraphobia.

In the current application, the investigators propose a five-year study to show the acute and longer-term effects of DCS augmentation of exposure-based CBT relative to placebo augmentation. This study is noteworthy for the use of a brief treatment strategy that has been shown to be successful in previous trials (e.g., Clark et al., 1999; Roy-Byrne et al., 2005) and has served as the basis for the DCS augmentation effect seen in a pilot study for this application. By demonstrating that DCS can enhance the results of even a brief treatment strategy, the investigators are seeking to validate an approach that fits well with the practice limitations and applications of CBT in effectiveness studies (e.g., Katon et al., 2006; Roy-Byrne et al. 2005). Furthermore, by studying the genetic predictors of the overall response to CBT, and DCS augmentation in particular, the investigators hope to further elucidate the nature of DCS augmentation and the selection of particularly responsive subgroups of patients in need. This agenda is in accords with "the ultimate goal of personalized therapy: identifying individual patterns of pathophysiology that indicate which pharmacological or behavioral treatment will be most useful for any individual patient" (Anderson & Insel, 2006, p. 320).

The study design is a double blind, randomized, controlled, trial conducted at three treatment sites. Patient with panic disorder will randomly receive DCS or placebo 1 hour prior to sessions 3-5 of a 5-session CBT protocol that includes 2 additional booster sessions over the course of follow-up. Patients will be enrolled over 5 years with the identical treatment protocol followed at each of the sites. Sites will nonetheless differ with respect to study management and analysis procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients > 18 years of age with a primary psychiatric diagnosis of panic disorder with or without agoraphobia
* CGI-severity score of 4 or higher
* Physical examination and laboratory findings without clinically significant abnormalities
* Off concurrent psychotropic medication for at least 2 weeks prior to initiation of randomized treatment, OR stable on current medication for a minimum of 6 weeks and willing to maintain a stable dose
* Willingness and ability to comply with the requirements of the study protocol

Exclusion Criteria:

* Agoraphobia sufficiently severe as to limit patient's ability to travel to and participate in weekly sessions Posttraumatic stress disorder, substance use disorder, eating disorder, or organic mental disorder within the past 6 months
* Lifetime history of psychotic disorder, bipolar disorder, or developmental disorder
* Significant suicidal ideation or suicidal behaviors within the past 6 months
* Significant personality dysfunction likely to interfere with study participation
* Serious medical illness or instability for which hospitalization may be likely within the next year
* Patients with a current or past history of seizures (other than febrile seizures in childhood)
* Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception
* Concurrent psychotherapy initiated within 3 months of baseline, or ongoing psychotherapy of any duration directed specifically toward treatment of the panic disorder other than general supportive therapy initiated at least 3 months prior to study
* Prior adequate trial of CBT for panic disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Otto, PhD, Study Chair — Boston University; David F Tolin, PhD, Principal Investigator — Institute of Living; Mark H Pollack, MD, Principal Investigator — Rush University Medical Center
Locations (4):
- United States (4):
  - Institute of Living, Hartford, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Otto MW, Pollack MH, Dowd SM, Hofmann SG, Pearlson G, Szuhany KL, Gueorguieva R, Krystal JH, Simon NM, Tolin DF. RANDOMIZED TRIAL OF D-CYCLOSERINE ENHANCEMENT OF COGNITIVE-BEHAVIORAL THERAPY FOR PANIC DISORDER. Depress Anxiety. 2016 Aug;33(8):737-45. doi: 10.1002/da.22531. Epub 2016 Jun 17. PMID 27315514

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled at Boston University (n = 68), the Institute of Living in Hartford, Connecticut (n = 59), and a combined site of Massachusetts General Hospital and Rush University Medical Center (n = 53). Results presented here are for all sites.
Pre-assignment Details: 293 individuals completed baseline evaluations. Of these, 98 were deemed ineligible (e.g., other primary diagnosis, medication exclusion) at the initial screening visit. An additional 15 participants were not randomized due to withdrawal (n = 4), lost to follow-up (n = 10), and changes to medication (n = 1). 180 participants were randomized.
Period: Overall Study
Arm/Group | D-cycloserine | Placebo
Started (98 participants were deemed ineligible at baseline and 15 others were not randomized.) | 88 | 92
Completed (All randomized participants (n = 180) were included in data analysis.) | 82 | 75
Not Completed | 6 | 17
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 2 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine | Placebo | Total
Number analyzed (Participants) | 88 | 92 | 180
Age, Categorical [Count of Participants; unit: Participants] — Population: Complete demographic information was collected for 178 participants. Some or all demographic information is missing for the remaining 2 participants.
  Participants
    number analyzed (Participants) | 87 | 91 | 178
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 85 | 90 | 175
    >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Measure Analysis Population Description: Complete demographic information was collected for 178 participants. Some or all demographic information is missing for the remaining 2 participants.
  Years
    number analyzed (Participants) | 87 | 91 | 178
    (all) | 35.75 (11.59) | 35.18 (12.84) | 35.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Complete demographic information was collected for 178 participants. Some or all demographic information is missing for the remaining 2 participants.
  Participants
    Female | 49 | 58 | 107
    Male | 39 | 34 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Complete demographic information was collected for 178 participants. Some or all demographic information is missing for the remaining 2 participants (with 1 subject missing ethnicity, and 1 subject missing race due to confused reporting of these terms).
  Participants
    Hispanic or Latino | 7 | 12 | 19
    Not Hispanic or Latino | 81 | 79 | 160
    Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Complete demographic information was collected for 178 participants. Some or all demographic information is missing for the remaining 2 participants (with 1 subject missing ethnicity, and 1 subject missing race due to confused reporting of these terms).
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 5 | 9
    White | 81 | 85 | 166
    More than one race | 1 | 1 | 2
    Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: Complete demographic information was collected for 178 participants. Some or all demographic information is missing for the remaining 2 participants.
  Participants
    United States: Boston University | 33 | 35 | 68
    United States: Institute of Living in Hartford, Connecticut | 29 | 30 | 59
    United States: Massachusetts General Hospital/Rush | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Panic Disorder Severity Scale (PDSS)
Description: The percent change in PDSS score from baseline to the relevant assessment points is the continuous primary outcome measure. The PDSS consists of seven items, each rated on a 0 to 4 scale (0 denoting none, and higher ratings reflecting greater degrees of symptom severity; for a possible range in scores from 0 to 28). In the tabular data below we present the total scores (sum of items).
Time Frame: baseline, mid-TX, post-TX, follow-up visits 1-4
Population: Seventeen subjects out of 92 (five during treatment and 12 during follow-up, 20% total) in the control group compared to six out of 88 (four during treatment and two during follow-up, 10% total) in the DCS group dropped out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 88 | 92
units on a scale
  Baseline | 13.30 (4.50) | 13.37 (3.39)
  TX Midpoint: number analyzed (Participants) | 87 | 91
  TX Midpoint | 7.98 (3.92) | 8.32 (4.19)
  TX Endpoint: number analyzed (Participants) | 84 | 87
  TX Endpoint | 5.30 (3.52) | 6.43 (4.63)
  Follow-Up 1: number analyzed (Participants) | 83 | 81
  Follow-Up 1 | 4.76 (3.82) | 5.84 (4.36)
  Follow-Up 2: number analyzed (Participants) | 85 | 83
  Follow-Up 2 | 4.38 (3.50) | 4.53 (4.03)
  Follow-Up 3: number analyzed (Participants) | 83 | 79
  Follow-Up 3 | 4.46 (3.76) | 4.35 (4.07)
  Follow-Up 4: number analyzed (Participants) | 82 | 75
  Follow-Up 4 | 3.85 (3.44) | 3.45 (3.78)

2. Primary Outcome: Remission Status
Description: Remission status will be used as the primary categorical outcome variable. The CGI-S was used in determining whether patients met the "CGI-S of 1 or 2" component of the "remission status" criteria (i.e., zero panic attacks and CGI-S of 1 or 2 at endpoint). No values are missing because remission must be confirmed; missing status is assigned to disorder status. Hence results are for the full randomized sample.
Time Frame: Pre-treatment, Post-Treatment, and each follow-up sessions
Population: Full sample of 180 randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 88 | 92
Participants
  Mid-Treatment | 8 | 4
  Tx Endpoint | 23 | 26
  Follow Up-1 | 42 | 34
  Follow Up-2 | 47 | 49
  Follow Up-3 | 48 | 52
  Follow Up-4 | 54 | 63

3. Secondary Outcome: Depression Severity
Description: Depression severity was assessed with the MADRS, with scores ranging from 0 to 60. Higher scores indicate greater depression.
Time Frame: Baseline, Tx Endpoint, Each of 4 follow-up assessments
Population: Randomized participants with panic disorder
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 88 | 92
units on a scale
  Baseline | 11.4 (8.5) | 11.4 (8.8)
  Treatment Endpoint: number analyzed (Participants) | 84 | 87
  Treatment Endpoint | 6.9 (6.8) | 7.8 (8.5)
  Follow Up-1: number analyzed (Participants) | 81 | 83
  Follow Up-1 | 7.5 (7.5) | 8.1 (8.3)
  Follow Up-2: number analyzed (Participants) | 85 | 83
  Follow Up-2 | 7.4 (7.4) | 7.1 (8.4)
  Follow Up-3: number analyzed (Participants) | 83 | 78
  Follow Up-3 | 7.0 (7.6) | 6.1 (7.8)
  Follow Up-4: number analyzed (Participants) | 82 | 75
  Follow Up-4 | 6.1 (6.5) | 6.7 (6.7)

4. Secondary Outcome: Quality of Life Ratings
Description: Quality of life as assessed by the Q-LES-Q. Scores range from 14-70 for total raw score, higher scores indicate higher quality of life ratings.
Time Frame: Baseline, Tx Endpoint, Each of 4 follow-up assessments
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 88 | 92
units on a scale
  Baseline | 47.2 (9.3) | 47.1 (9.9)
  TX - Endpoint: number analyzed (Participants) | 84 | 86
  TX - Endpoint | 54.4 (7.7) | 52.7 (9.2)
  Follow Up-1: number analyzed (Participants) | 83 | 81
  Follow Up-1 | 53.9 (7.8) | 52.2 (9.4)
  Follow Up-2: number analyzed (Participants) | 85 | 82
  Follow Up-2 | 54.3 (7.8) | 53.4 (9.2)
  Follow Up-3: number analyzed (Participants) | 83 | 78
  Follow Up-3 | 54.6 (8.4) | 55.1 (8.6)
  Follow Up-4: number analyzed (Participants) | 82 | 75
  Follow Up-4 | 55.6 (7.9) | 54.7 (8.7)

5. Secondary Outcome: Role Functioning
Description: LIFE-RIFT. For this clinician-rated measure, total scores range from 0 to 20, with higher scores indicating greater impairment
Time Frame: Baseline, Tx Endpoint, Each of 4 follow-up assessments
Population: Randomized sample
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 88 | 92
units on a scale
  Baseline | 9.7 (3.5) | 9.8 (3.0)
  TX - Endpoint: number analyzed (Participants) | 84 | 87
  TX - Endpoint | 7.7 (2.8) | 8.2 (2.8)
  Follow Up-1: number analyzed (Participants) | 83 | 81
  Follow Up-1 | 7.6 (2.8) | 7.9 (2.7)
  Follow Up-2: number analyzed (Participants) | 85 | 83
  Follow Up-2 | 7.4 (2.8) | 7.5 (2.6)
  Follow Up-3: number analyzed (Participants) | 83 | 78
  Follow Up-3 | 7.2 (2.7) | 6.8 (2.4)
  Follow Up-4: number analyzed (Participants) | 82 | 75
  Follow Up-4 | 7.1 (2.7) | 7.2 (2.6)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and elicited by open questioning of the study clinician, assessing adverse events occurring over the last hour as well as during the week following the last dose of DCS. AEs and SAEs were informally assessed up to the 6-month follow-up.
Arm/Group | D-cycloserine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/92
Serious Adverse Events (participants affected / at risk) | 1/88 | 1/92
Other Adverse Events (participants affected / at risk) | 17/88 | 18/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine (N=88) | Placebo (N=92)
Pancreatitis (Endocrine disorders) | 1 (1) | 0 (0) — One participant was hospitalized for pancreatitis and released the following morning. Follow-up care included additional testing to determine best course of action. This event was judged to be unrelated to the study procedures.
Appendicitis (Endocrine disorders) | 0 (0) | 1 (1) — One participant was hospitalized for the treatment of appendicitis. At the time, the participant was in the active phase of the study. This event was judged to be unrelated to study procedures.
Kidney Infection (Renal and urinary disorders) | 0 (0) | 0 (0) — A participant was hospitalized for a kidney infection for one day. This event happened prior to randomization of the study drug. The investigators judged this event to be unrelated to the study procedures.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | D-cycloserine (N=88) | Placebo (N=92)
Nausea/vomiting (Gastrointestinal disorders) | 6 | 7
Gastrointestinal distress (Gastrointestinal disorders) | 2 | 3
Headache (General disorders) | 4 | 3
Fatigue (General disorders) | 11 | 3
Sedation (General disorders) | 5 | 3
Jitteriness/tremor (General disorders) | 3 | 1
Agitation/restlessness (General disorders) | 2 | 0
Dizziness/lightheadedness (General disorders) | 5 | 10
Anxiety/panic (Psychiatric disorders) | 2 | 0
Impaired concentration (Psychiatric disorders) | 1 | 1
Dry mouth (General disorders) | 4 | 1
Blurred vision (Eye disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 2 | 0
Paresthesias (General disorders) | 1 | 4
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Itching (Skin and subcutaneous tissue disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Derealization (Psychiatric disorders) | 1 | 1
Menstrual irregularity (Reproductive system and breast disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The investigators did not systematically collect fear estimates across exposure and are therefore unable to examine this factor as a moderator.

Unexpected site effects were observed for several of our outcome variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No